CLINICAL TRIAL: NCT06984588
Title: A Phase II/III, Randomized, Multicenter, Open-Label Study to Compare Uliledlimab Combined With Toripalimab, Toripalimab Monotherapy, and Pembrolizumab Monotherapy in Patients With Previously Untreated Locally Advanced Unresectable or Metastatic PD-L1- and CD73- Selected Non-Small Cell Lung Cancer
Brief Title: A Study to Compare Uliledlimab Combined With Toripalimab, Toripalimab Monotherapy, and Pembrolizumab Monotherapy in Patients With Previously Untreated Locally Advanced Unresectable or Metastatic PD-L1- and CD73- Selected Non-Small Cell Lung Cancer
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: TJ Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TJ004309LUC301
Record Dates: First submitted 2025-04-22; First posted 2025-05-22 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — toripalimab; pembrolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental)
  Interventions: Drug: Uliledlimab; Drug: Toripalimab
- Group B (Active Comparator)
  Interventions: Drug: Pembrolizumab
- Group C (Sham Comparator)
  Interventions: Drug: Toripalimab

INTERVENTIONS:
Drug: Uliledlimab — 30 mg/kg, administered on Days 1 and 8 of Cycle 1 (C1D1 and C1D8), then once every 3 weeks (Q3W) starting from C2D1,
  Arms: Group A
Drug: Toripalimab — 240 mg on Day 1, once every 3 weeks (Q3W)
  Arms: Group A; Group C
Drug: Pembrolizumab — 200 mg on Day 1, once every 3 weeks (Q3W)
  Arms: Group B

SUMMARY:
This is a Phase II/III, randomized, open-label, active-controlled, multicenter study to compare intravenous uliledlimab combined with toripalimab, toripalimab monotherapy, and pembrolizumab monotherapy in patients with previously untreated locally advanced unresectable or metastatic PD-L1-positive (tumor proportion score [TPS] ≥ 1%) and CD73-positive (TC/IC > 30%; TC/IC defined as the higher of either the proportion of CD73-positive tumor cells or the proportion of CD73-positive immune cells at any intensity [IHC1+ or above]) NSCLC who are not suitable for targeted therapies such as EGFR, ALK, etc.

The number of enrolled subjects with PD-L1 TPS ≥ 50% will be limited to approximately 60% of the total sample size to reflect the natural prevalence of advanced NSCLC.

Patients who have received adjuvant or neoadjuvant therapy other than immune checkpoint inhibitor treatments are allowed to participate in this study, provided that such treatments have been completed at least 12 months prior to the occurrence of recurrence or metastasis.

During the screening period, tumor samples will be collected in advance and tested by the central laboratory for PD-L1 expression levels using the PD-L1 IHC 22C3 pharmDx assay and CD73 expression levels using the CD73 antibody assay (immunohistochemistry). Previous PD-L1 testing results obtained using the PD-L1 IHC 22C3 pharmDx assay will be accepted. Patients with PD-L1 positive expression (TPS ≥ 1%) and high CD73 expression (TC/IC > 30%) will meet the inclusion criteria.

Patients who do not meet the eligibility criteria as judged by the investigator may be re-screened once.

Patients with non-squamous NSCLC will be required to confirm the absence of EGFR-sensitive mutations or ALK fusion; patients with unknown EGFR and ALK expression status will be required to undergo testing and provide clinical laboratory test results prior to study enrollment, and may be enrolled after relevant driver gene mutations are ruled out. Meanwhile, patients with other definite actionable driver gene alterations (such as: ROS1 fusions, RET fusions, NTRK1/2/3 fusions, BRAF V600E mutations, MET14 exon skipping mutations, etc.) will be excluded from this study. Controversial cases with actionable gene mutations will be submitted to the study expert panel for joint decision.

This study includes Phase II and Phase III stages. Approximately 150 subjects will be enrolled in the Phase II stage. Based on the evaluation of the efficacy, safety, PK, and PD results of the Phase II study, a decision will be made on whether to proceed to the Phase III study. Approximately 300 subjects will be enrolled in the Phase III stage.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥ 18 years at the time of signing the ICF
2. Patients with histologically or cytologically confirmed stage IIIB, IIIC, or IV NSCLC (according to the American Joint Committee on Cancer Staging System, 8th edition) who are not suitable for radical surgery and/or radiotherapy (with or without chemotherapy).
3. Patients who have not received prior systemic therapy for their locally advanced or metastatic diseases.
4. Patients with measurable lesions as assessed by the investigator at the study site based on RECIST v1.1. Target lesions located in a previously irradiated region will be considered measurable only if there is documented evidence of disease progression
5. Patients with non-squamous NSCLC who are confirmed to have no EGFR-sensitive mutations or ALK fusions.
6. Patients with PD-L1 TPS ≥ 1% and CD73 TC/IC > 30% (IHC1+ or higher). It will be tested by the central laboratory for PD-L1 expression levels using the PD-L1 IHC 22C3 pharmDx assay, and CD73 expression levels using the CD73 antibody assay.
7. Patients with a life expectancy of at least 3 months.
8. Patients with Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
9. Patients with adequate organ function
10. Patients with negative HIV testing at screening.
11. Patients with negative hepatitis B virus surface antigen (HBsAg) or inactive hepatitis B (HBsAg positive with HBV-DNA copy number ≤ ULN, ALT ≤ ULN, and no treatment is required in the investigator's opinion) at screening.
12. Patients with negative hepatitis C virus (HCV) antibody at screening, or positive HCV antibody and negative HCV RNA at screening.
13. For women of childbearing potential: A urine or serum pregnancy test must be negative within 72 hours prior to the first dose of study drug. If the urine pregnancy test result is positive or cannot be confirmed as negative, a serum pregnancy test should be performed.
14. For male subjects with female partners of childbearing potential: They must agree to use an effective method of contraception from the first dose of study drug to 180 days after the last dose of study drug.Male subjects with pregnant partners will be required to agree to use condoms; pregnant partners will not be required to use additional methods of contraception.
15. Patients who voluntarily agree to participate in the study and sign a written ICF

Exclusion Criteria:

1. Patients who are currently pregnant, breastfeeding, or planning to conceive or give birth within the expected duration of this study.
2. Patients previously treated with immune checkpoint inhibitors.
3. Patients who are receiving or have completed systemic immune agonist therapy (including but not limited to: interferon and interleukin-2) within 4 weeks prior to the first dose or 5 drug elimination half-lives (whichever is longer).
4. Patients who have received oral or intravenous antibiotic therapy within 2 weeks prior to starting study treatment, except for prophylactic use.
5. Patients who have undergone major surgery within 4 weeks prior to starting study treatment, except for diagnostic surgery.
6. Patients who have received a live attenuated vaccine within 30 days prior to starting study treatment. Seasonal influenza vaccines that do not contain live viruses are permitted.
7. Patients who are currently participating in another clinical trial and receiving study treatment, or who have participated in a clinical trial and received investigational drug or device treatment within 4 weeks prior to enrollment.
8. Patients who have received any anti-tumor therapeutic agents containing traditional Chinese medicine ingredients within 4 weeks prior to starting study treatment.
9. Patients who have previously received an allogeneic tissue/organ transplant.
10. Patients who are expected to require any other form of anti-tumor therapy during the course of the study.
11. Patients who are receiving radiotherapy, with the exception of: 1) local radiotherapy for brain lesions, refer to exclusion criterion 22; 2) palliative radiation for bone metastases, provided that it is completed at least 7 days prior to randomization and the patient's condition is stable.
12. Patients with angina, myocardial infarction, symptomatic congestive heart failure, cerebrovascular accident, transient ischemic attack, arterial embolism, unstable arrhythmia, pulmonary embolism, or treatment with percutaneous transluminal coronary angioplasty or coronary artery bypass grafting within 6 months prior to study treatment.
13. Patients with hypertension (defined as systolic blood pressure > 150 mmHg or diastolic blood pressure > 90 mmHg) or CTCAE Grade ≥2 hypotension.
14. Patients with uncontrolled or symptomatic hypercalcaemia (> 1.5 mmol/L ionized calcium or calcium > 12 mg/dL or corrected serum calcium > ULN).
15. Patients with known previous malignancies other than NSCLC, except for those who have received radical therapy, have no evidence of disease recurrence within 5 years, and are assessed by the investigator to be at low risk of recurrence.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2024-03-28 (Actual); Primary Completion 2028-08-05 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | From the date of randomization to the date of first documented disease progression (assessed by a blinded independent central review [BICR] according to RECIST v1.1) or death from any cause, whichever occurs first,assessed up to 6 months

CONTACTS AND LOCATIONS:
Locations (64):
- China (64):
  - Anyang Tumour Hospital, Anyang
  - Beijing Chest Hospital, Capital Medical University, Beijing
  - Bejing Chao-Yang Hospital, Capital Medical University, Beijing
  - The First Affiliated Hospital of Bengbu Medical University, Bengbu
  - Binzhou Medical University Hospital, Binzhou
  - The Third Xiangya Hospital of Central South University, Changsha
  - Xiangya Hospital of Central South University, Changsha
  - Army characteristic Hospital Center( Daping Hospital of the Third Military Medical University), Chongqing
  - Chongqing University Cancer Hospital, Chongqing
  - Chongqing University Three Gorges Hospital, Chongqing
  - The People's Hospital of Dongguan, Dongguan
  - The first people's hospital of Foshan, Foshan
  - First Affiliated Hospital of Gannan Meidcal University, Ganzhou
  - Ganzhou People's Hospital, Ganzhou
  - Guangdong Provincial People's Hospital, Guangzhou
  - Guizhou Provincial People's Hospital, Guiyang
  - The Second Affiliated Hospital of Hainan Medical University, Haikou
  - Harbin Medical university cancer hospital, Ha’erbin
  - Anhui provincial cancer hospital, Hefei
  - The First Affiliated Hospital of Anhui Medical University, Hefei
  - Jiamusi Tumour Hospital, Jiamusi
  - Jiangmen Central hospital, Jiangmen
  - Jinan Central Hospital, Jinan
  - Affiliated Hospital of Jining Medical University, Jining
  - Linyi People's Hospital, Linyi
  - Lishui Central Hospital, Lishui
  - Liuzhou Central Hospital, Liuchow
  - Longyan First Hospital, Longyan
  - Jiangxi Cancer Hospital, Nanchang
  - The First Affiliated Hospital Of Nanchang University, Nanchang
  - Nanchong Central Hospital, Nanchong
  - Jiangsu Province Hospital, Nanjing
  - Guangxi Medical University Cancer Hospital, Nanning
  - The First Affiliated Hospital of Guangxi Medical University, Nanning
  - Nantong Tumor Hospital, Nantong
  - Nanyang Cenreal Hospital, Nanyang
  - The Second People's Hospital of Neijiang, Neijiang
  - Qingdao Central Hospital, Qingdao
  - The First People's Hospital Of Qujing, Qujing
  - Yuebei People's Hospital, Shaoguan
  - China Shenyang the Tenth People's Hospital(China Shenyang Chest Hospital), Shenyang
  - The Fourth Hospital Of Hebei Medical University, Shijia Zhuang
  - Suining Central Hospital, Suining
  - First Hospital of Shanxi Medical University, Taiyuan
  - Taizhou Hospital of Zhejiang Province, Taizhou
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin
  - Union Hospital affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - The Second Affiliated Hospital Of Xi'an Jiaotong University, Xi'an
  - Xi'an Chest Hospital, Xi'an
  - Fujian Provincial Cancer Hospital, Xiamen
  - The First Affiliated Hospital Of Xiamen University, Xiamen
  - The Second Affiliated Hospital of Xiamen Medical College, Xiamen
  - Xiangyang Central Hospital, Xiangyang
  - Northern Jiangsu People's Hospital, Yangzhou
  - The Second People's Hospital Of Yibin, Yibin
  - Yichang Central People's Hospital, Yichang
  - Shanxi Yuncheng Central hospital, Yuncheng
  - The First Affiliated Hospital Of Henan University Of Science & Technology, Zhengzhou
  - The First Affiliated Hospital Of Zhengzhou University, Zhengzhou
  - Zhoukou Central hospital, Zhoukou
  - Zhujiang hospital of Southern Medical University, Zhujiang
  - Zibo Municipal Hospital, Zibo
  - The first people's hospital of Zunyi, Zunyi

IPD SHARING:
Plan to Share IPD: No